CLINICAL TRIAL: NCT03844529
Title: Evaluation of Collagen Dermal Filler With Lidocaine for the Correction of Nasolabial Folds: a Prospective, Randomized, Active-controlled, Double Blinded, Multicenter Clinical Trial
Brief Title: Evaluation of Collagen Dermal Filler With Lidocaine for the Correction of Nasolabial Folds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Tri-Service General Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201809007DSA
Record Dates: First submitted 2019-01-31; First posted 2019-02-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-01

CONDITIONS: Nasolabial Fold

STUDY DESIGN:
Intervention Model Description: 240 subjects will be recruited in total, and each hospital will recruit 60~120 subjects.
Who Masked: Participant, Investigator
Masking Description: This is a double blinded( blinded evaluator and subject) clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sunmax FULLSGEN with Lidocaine (Experimental): A subject would only receive single injection treatment(day 1) using Sunmax FULLSGEN , and there would be 6 follow-up visits at 4th, 12th, 24th, 36th and 52nd week after injection treatment.
  Interventions: Device: Sunmax FULLSGEN with Lidocaine
- Sumax FACIALGAIN collagen Implant with Lidocaine (Active Comparator): A subject would only receive single injection treatment(day 1) using Sumax FACIALGAIN collagen Implant with Lidocaine, and there would be 6 follow-up visits at 4th, 12th, 24th, 36th and 52nd week after injection treatment.
  Interventions: Device: Sunmax FULLSGEN with Lidocaine

INTERVENTIONS:
Device: Sunmax FULLSGEN with Lidocaine — Subject who voluntarily sign the informed consent form (day -14~1) will be randomly assigned to investigational or control group and have intradermal allergy test. After the injection treatment by randomly choosing the device, every subject would have 6 follow-up visits.
  Other Names: Sumax FACIALGAIN collagen Implant with Lidocaine

SUMMARY:
Evaluation the efficacy and safety of collagen dermal filler with lidocaine using in the middle to deep dermis for the correction of nasolabial folds.

DETAILED DESCRIPTION:
This is a prospective, randomized, active-controlled, double blinded (blinded evaluator and subject), multicenter clinical trial, which will be performed in Tri-Service General Hospital, Linkou ChangGung Memorial Hospital and National Taiwan University Hospital. These hospitals will recruit subjects in a competitive way. 240 subjects will be recruited in total, and each hospital will recruit 60~120 subjects. The expected execution period is 2018/10~2021/06. Subjects will be randomly assigned to receive the investigational device "Sumax FULLSGEN with Lidocaine" or controlled device "Sumax FACIALGAIN collagen Implant with Lidocaine" in 1:1 ratio. These devices will be processed to keep subjects and evaluators blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral defects in the nasolabial folds with grades 3 or 4 on the Wrinkle Severity Rating Scale (WSRS).
2. Male or female aged 20 ~ 65-year-old.
3. Willingness to receive wrinkle augment treatment.
4. Willingness to avoid other facial beauty therapy during this clinical trial.
5. Healthy facial skin condition, and not have any disorder that can interfere the assessment of skin aging, e.g. facial nerve disorders.
6. All the enrolled subjects should sign and date the informed consent form before this trial starts.

Exclusion Criteria:

1. Known history of anaphylactoid reaction and other auto-immune diseases.
2. Known history of allergies to collagen, or those who are allergic to the control or investigational device after the verification of intradermal allergy test.
3. Known history of allergies to lidocaine.
4. Known coagulation disorders.
5. Females who have positive pregnancy test at screening, plan a pregnancy, breastfeeding, and those who are unable to take contraception method.
6. Subjects with local infection, severity skin disease, inflammation or related symptoms on the nasolabial folds. Or with keloid (hypertrophic scar).
7. Subjects with severe cardiac, renal, hepatic, or respiratory diseases.
8. Subjects with clinically diagnosed mental illness.
9. According to American National Institute of Health standards, those who meet the criteria of Alcohol Use Disorder.
10. Subjects take immunosuppressive drugs, chemotherapy, or systemic steroids (i.e. oral or injection) within 12 weeks before screening.
11. Subjects take anticoagulant treatment or NSAIDs within 1 week before screening.
12. Subjects have permanent implants in the nasolabial folds area.
13. Subjects have nasolabial folds augment treatment such as autologous fat, hyaluronic acid or collagen filler implant within 52 weeks before screening.
14. Subjects have nasolabial fold correctional procedure or treatment such as botulinum toxin injection, chemical peeling, laser at dermis or plastic surgery.
15. Subjects unable to comply the scheduled follow-up.
16. Subjects participate other clinical trials within 12 weeks before screening (trials only with questionnaire or specimen collection are exemption).
17. Subjects who are not eligible for this trial based on the judgment of investigators.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
WSRS score evaluation | 24th week. Using the 5-grade Wrinkle Severity Rating Scale (WSRS) to evaluate wrinkle, and score 5 is the worst one.
  24th week response rate will be calculated according to WSRS score assessed by the evaluators Subtract the subject's WSRS baseline score from the Xth week after injection as improved score.

SECONDARY OUTCOMES:
WSRS score evaluation within 4 time point as assessed by the evaluators | 4th, 12th, 36th and 52nd week week. Using the 5-grade Wrinkle Severity Rating Scale (WSRS) to evaluate wrinkle, and score 5 is the worst one.
  WSRS response rate at 4th, 12th, 36th and 52nd week as assessed by the evaluators
GAIS score at specific week as assessed by the subject | 4th, 12th, 24th, 36th and 52nd week. Global Aesthetic Improvement Scale (GAIS) is scored 5 level of improvement. Score 5 is the worst value.
  GAIS score at 4th, 12th, 24th, 36th and 52nd week as assessed by the subject
GAIS score at specific week as assessed by the evaluators | 4th, 12th, 24th, 36th and 52nd week. Global Aesthetic Improvement Scale (GAIS) is scored 5 level of improvement. Score 5 is the worst value.
  GAIS score at 4th, 12th, 24th, 36th and 52nd week as assessed by the evaluators
VAS score evaluation | 30 minutes. Double-sided print or photocopy the next 2 diagrams ensuring that the lines are exactly 10 cm in length and superimposed.
  VAS score within 30 mins after injection as assessed by the subject
TPS score evaluation | 30 minutes. The score is evaluated by thermometer pain scale, and the scale is 0-10. 0 stands for on pain, and 10 stands for worst possible pain.
  TPS score within 30 mins after injection as assessed by the investigator

OTHER OUTCOMES:
Safety Endpoint (Evaluation of laboratory inspection values.) | One year. Number of participants with abnormal laboratory values and/or adverse events that are related to treatment.
  Evaluation of laboratory inspection values.
Safety Endpoint (Evaluation of the percentage of AE and AR) | One year. Number of participants with AE divided by number of participants with AR is the percentage of AE and AR.
  Evaluation of the percentage of AE and AR

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No